CLINICAL TRIAL: NCT06479954
Title: ELREXFIO SPECIAL INVESTIGATION- INVESTIGATION ON LONG-TERM TREATMENT -
Brief Title: Non Interventional Study to Investigate the Safety and Effectiveness in Patients With Relapsed and Refractory Multiple Myeloma Treated With Elranatamab Under the Actual Use.
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C1071010
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Relapsed and Refractory Multiple Myeloma (RRMM)
Keywords: RRMM
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To investigate the safety and efficacy in patients with relapsed and refractory multiple myeloma treated with elranatamab under the actual use.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and efficacy in patients with relapsed and refractory multiple myeloma (RRMM) treated with elranatamab under the actual use.

* Primary objective: Confirm whether the onset status (the number of patients, incidence, grade, seriousness, timing of onset, duration, treatment and outcome) of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) is comparable to that in the clinical studies and whether adverse reactions were appropriately treated.
* Secondary objective: Confirm the onset status of any adverse reaction (including unknown adverse reaction) to long-term treatment with elranatamab and the overall response (ORR) as efficacy assessment and evaluate them in terms of benefit-risk.

Conditions for approval; Because of the extremely limited number of patients treated in Japanese clinical studies, a drug use investigation in all patients should be conducted to understand the background information of patients on elranatamab, early collect data on the safety and efficacy of elranatamab, and take measures necessary for the proper use of elranatamab until the data of a certain number of patients are accumulated.

ELIGIBILITY:
Inclusion Criteria:

Patients who have received at least one dose of elranatamab.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All of the patients who satisfy all of the registration criteria in all the institutions to which elranatamab is delivered based on the conditions for approval are subject to this study.
  registration criteria ;Patients who have received at least one dose of elranatamab.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of CRS events in adverse drug reaction | up to 52 weeks
  An adverse drug reaction (ADR) in cytokine release syndrome (CRS) was any untoward medical occurrence attributed to Elrexfo in a participant who received this drug. A serious ADR (SADR) was an ADR resulting in any of the following out comes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Elrefxio was assessed by the physician.
Incidence of ICANS events in adverse drug reaction | up to 52 weeks
  An adverse drug reaction (ADR) in immune effector cell-associated neurotoxicity syndrome (ICANS) was any untoward medical occurrence attributed to Elrexfo in a participant who received this drug. A serious ADR (SADR) was an ADR resulting in any of the following out comes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Elrefxio was assessed by the physician.

SECONDARY OUTCOMES:
Proportion of patients with objective response rate (ORR) | up to 52 weeks
  Defined as stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR)
Incidence of other adverse drug reactions (ADRs) | up to 52 weeks
  An adverse drug reaction (ADR) was any untoward medical occurrence attributed to Elrexfo in a participant who received this drug. A serious ADR (SADR) was an ADR resulting in any of the following out comes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to Elrefxio was assessed by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1071010